CLINICAL TRIAL: NCT04504903
Title: Work as a Determinant of Health: A Pragmatic Trial of Enhanced Cognitive Behavioral Therapy to Bolster Competitive Work and Wellness in Veterans With Serious Mental Illness (WORKWELL)
Brief Title: Cognitive Behavioral Therapy to Improve Work and Wellness in Veterans With Mental Illness
Acronym: WORKWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 19-176
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Posttraumatic Stress Disorders
Keywords: Rehabilitation, Vocational
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Unemployed participants with serious mental illness will be randomized to receive group-based cognitive behavioral therapy geared toward improving competitive work outcomes or a time and format matched psychoeducation intervention
Who Masked: Outcomes Assessor
Masking Description: Research personnel conducting outcomes assessments will be blinded to condition assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy For Work Success (CBTw) (Experimental): Veterans will participate in 12 weekly group sessions to discuss thoughts, feelings, and behaviors that promote work success in the community
  Interventions: Behavioral: Cognitive Behavioral Therapy For Work Success (CBTw)
- Psychoeducation (Active Comparator): Veterans in the control group will participate in 12 weekly group sessions in which they will learn more about their mental health conditions.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy For Work Success (CBTw) — Veterans will go to 12 weekly group sessions and will learn healthy thinking about work, positive behavioral coping related to work, and will form a work success plan based on their work goals.
  Arms: Cognitive Behavioral Therapy For Work Success (CBTw)
Behavioral: Psychoeducation — Veterans will go to 12 weekly group sessions and will learn more information about their mental health conditions. Psychoeducation modules are from the Illness Management and Recovery program.
  Arms: Psychoeducation

SUMMARY:
Vocational instability in Veterans with serious mental illness (SMI) is pervasive, costly, and harmful. Over 75% of Veterans with SMI are unemployed, resulting in economic difficulties and trouble meeting basic needs. Overall, among adults with depression, work dysfunction results in a 36 to 51 billion dollar loss annually. Unemployed Veterans with SMI also suffer major health consequences, including a more severe course of illness and poor recovery over time, leading to increased inpatient and emergency service use. The WORKWELL study will synergistically address these deficits in health, recovery, and work functioning by testing the Cognitive Behavioral Therapy for Work Success (CBTw) intervention. Using a pragmatic design, this project will address work as a major social determinant of health and close the health disparity gap among people with SMI. Further, through promotion of work and healthy thinking, CBTw holds promise to reduce risk of suicide among vulnerable veterans with SMI.

DETAILED DESCRIPTION:
Project background: Work is a major social determinant of health. In people with serious mental illness (SMI), work is associated with better wellbeing, physical and mental health, quality of life, and may prevent the onset of disability. Among Veterans with SMI, work is a protective factor against suicide.

Most veterans with SMI are unemployed and suffer substantially worse health and recovery across key domains. Despite quality VHA vocational services, such as supported employment (SE), two-thirds or more of Veterans who receive these services experience work dysfunction. A probable explanation lies in unsolved cognitive and behavioral barriers, such as low work-related self-efficacy, ineffective coping skills, little hope that work is attainable, poor work motivation and sense of self.

The Cognitive Behavioral Therapy for Work Success (CBTw) intervention was designed to target these problems and augment VHA SE services to synergistically improve work, as well as health and recovery, in Veterans with SMI. In an open trial pilot, CBTw was associated with significant increases in hours worked and wages earned and the majority of CBTw participants became steady workers. Veterans also experienced improvements in symptoms, recovery, and quality of life.

Project goals: Using Hybrid 1 RCT design, this project will test the effects of CBTw on competitive work and health and recovery outcomes over a 12-month study period at 3 VA SE programs. Informed by the RE-AIM framework, an implementation evaluation will examine the success of using SE staff to deliver CBTw, barriers and facilitators to implementation, and strategies utilized.

Relevance to priorities: This project has high implementation potential and is responsive to the VHA priority regarding Health Equity, as it will address work functioning, an under studied social determinant of health. WORKWELL also holds promise to improve health and recovery outcomes among Veterans with SMI, another HSR&D area of emphasis. Lastly, this study is consistent with the goal of finding novel strategies toward suicide prevention among vulnerable Veteran groups, including those with SMI.

Objectives: Aim 1: Test the effects of CBTw + SE compared to a control of psychoeducation + SE on work. Hypotheses: Participants in the CBTw+ SE arm will work significantly more total weeks in competitive jobs (primary study outcome) and will be more likely to become steady workers.

Aim 2: Test the effects of CBTw + SE on health and recovery. Hypotheses: Participants in the CBTw + SE arm will have greater improvements on subjective recovery and health-related quality of life, and decreases in symptoms, suicidal ideation, and inpatient service utilization.

Aim 3: Guided by the RE-AIM implementation science framework, conduct an evaluation of the implementation of CBTw, including examination of the feasibility of using SE staff to deliver CBTw, and related barriers and facilitators. The objective is to spur future wide scale CBTw implementation.

Project Methods: WORKWELL is a pragmatic, Hybrid 1 design RCT. CBTw will be tested at 3 SE sites-Roudebush VA Medical Center, the Edward J. Hines VA Medical Center, and the VA St. Louis Health Care System. 276 unemployed Veterans with SMI will be randomly assigned to receive CBTw plus SE or a control of psychoeducation plus SE. Outcomes including total weeks worked in competitive jobs (primary), achievement of steady work, symptoms, recovery, health related quality of life, suicidal ideation, and service utilization will be assessed at posttreatment (12 weeks), 6 months (primary endpoint), and 9 months (to examine sustained effects). Primary work outcomes will be collected monthly over a 12-month period. CBTw implementation planning, training, and consultation will be provided. CBTw implementation (fidelity), barriers and facilitators to implementation, and other RE-AIM elements will be examined using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Unemployment, defined as no current participation in a competitive job
* A competitive work goal, which denotes a goal of a regular job in the community that pays at least minimum wage
* Presence of a serious mental illness including one or more of the following conditions:

  * major depression
  * bipolar disorders
  * schizophrenia
  * schizoaffective disorder
  * posttraumatic stress disorder (PTSD)
* Currently enrolled in and receiving VA vocational rehabilitation services

Exclusion Criteria:

* Previous participation in cognitive behavioral therapy intervention geared toward work
* Presence of a severe medical or cognitive impairment that will prevent participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Total weeks worked in competitive jobs change | baseline to 12 months
  Outcome measure will be mean number of weeks worked in competitive jobs. The primary endpoint is 6 months (primary comparison will be baseline to 6 months). Competitive jobs are regular jobs open to all that pay at least minimum wage. More total weeks worked in competitive jobs is indicative of a positive outcome.

SECONDARY OUTCOMES:
Achievement of steady competitive work change | baseline to 12 months
  Outcome measure of steady competitive work is defined as working at least 50% of the study period as assessed at the 12 month follow up period. Achievement of steady competitive work is a positive outcome.
Cross-Cutting Symptom Measure (CCSM) change | baseline to 9 months
  Outcome measure is a 23-item, Likert response (scored on a 0 to 4 scale), self-rated instrument that assesses 13 domains of psychiatric symptoms(e.g., depression, anxiety, psychosis, mania, sleep problems, self-harm, substance use, etc.) with higher scores indicating more severe total symptoms. Total scores range from 0 to 92.
12-item Short Form Survey (SF-12) change | baseline to 9 months
  The SF-12 outcome measure will assess health-related quality of life and is comprised of the Physical Component Summary (PCS) and Mental Component Summary (MCS). Total scores range from 0 to 100 with higher scores indicating higher health-related quality of life.
Scale for Suicidal Ideation change | baseline to 9 months
  Outcome measure is a 21-item interviewer rated measure of a continuum of suicidal ideation, including thoughts, attitudes, plans, and behaviors. Total scores range from 0 to 42 with higher scores indicating more suicidal ideation.
Recovery Assessment Scale change | baseline to 9 months
  Outcome measure is a 41 item self report survey that will assess subjective recovery attitudes. Total scores range from 41 to 164 with higher scores indicating higher levels of subjective recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Elizabeth Kukla, PhD MS BS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (3):
- United States (3):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the Research Service will consider requests for the final data sets underlying the publications to be provided to the public. The limited dataset will include de-identified data relevant to the specific request. Independent research groups can view relevant data to evaluate the extent that data sources support conclusions made by authors in published studies as well as observe additional emergent themes and view supplemental details that might not be included in publications.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available once the study team completes all analyses.
Access Criteria: The Research Service will evaluate individual requests.

REFERENCES:
- [Result] Kukla M, McGuire AB, Weber KC, Hatfield J, Henry N, Kulesza E, Rollins AL. An Investigation of Employment Hope as a Key Factor Influencing Perceptions of Subjective Recovery among Adults with Serious Mental Illness Seeking Community Work. Behav Sci (Basel). 2024 Mar 19;14(3):246. doi: 10.3390/bs14030246. PMID 38540549

DOCUMENTS (1):
  • Informed Consent Form (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04504903/ICF_000.pdf